CLINICAL TRIAL: NCT00008255
Title: Evaluation Of Uridine 5-Triphosphate Solution For Inhalation (UTP) As An Adjunct In The Diagnosis Of Lung Cancer By Sputum Cytology
Brief Title: INS316 in Diagnosing Lung Cancer in Patients With Untreated Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: MSKCC-00092; CDR0000068391 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1894
Record Dates: First submitted 2001-01-06; First posted 2004-05-05 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2001-05

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

INTERVENTIONS:
Drug: INS316
Other: sputum cytology

SUMMARY:
RATIONALE: Doctors can diagnose lung cancer by collecting mucus coughed up from the lungs and examining it under a microscope to look for cancer cells. Breathing in INS316 may make it easier for patients to cough up mucus.

PURPOSE: Randomized phase II trial to study the effectiveness of INS316 in helping to diagnose lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a cytological diagnosis of lung cancer can be obtained more frequently from sputum specimens following inhalation of INS316 compared to specimens obtained following placebo or compared to specimens spontaneously expectorated in patients with untreated lung cancer. II. Assess the relative sensitivity of sputum cytology in the diagnosis of lung malignancies in this patient population using these sputum collection regimens. III. Determine the quantity of macrophages in sputum of these patients using these techniques. IV. Determine if the number of macrophages in sputum obtained by these methods is predictive of the likelihood of obtaining a positive diagnosis of lung cancer in these patients. V. Determine the total amount of sputum expectorated from these patients using these techniques.

OUTLINE: This is a randomized, double-blind, placebo-controlled, cross-over, multicenter study. Patients are randomized to one of two arms, then cross-over to the other arm. Arm I: Patients receive INS316 by inhalation via a nebulizer. Sputum is collected throughout the dosing and for 1 hour post dosing. Arm II: Patients receive placebo in the same manner as INS136 in arm I. All patients receive both treatments. Patients receive the first dose no more than 7 days after screening, and the second dose 3 to 10 days after the first dose. Patients are followed 1 day after completion of the second treatment. The sputum samples are fixed and examined cytologically.

PROJECTED ACCRUAL: Approximately 100-130 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven primary lung cancer OR Presumptive diagnosis based on chest x-ray, CT scan, history, or symptoms No prior treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: FEV1 at least 35% predicted Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other comorbid condition that would preclude study

PRIOR CONCURRENT THERAPY: See Disease Characteristics At least 4 days since prior bronchoscopic examination or pulmonary fine needle aspiration biopsy At least 3 days since prior sputum induction No concurrent medication that would preclude study At least 30 days since prior investigational drugs (including INS316) or experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Korst, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States